CLINICAL TRIAL: NCT03188432
Title: A Phase II Trial Comparing Quality of Life After HIPEC in Patients With Stage IIIC and IV Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Hyperthermic Intraperitoneal Chemotherapy Trial Comparing Quality of Life in Patients With Stage IIIC-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00044434; NCI-2017-01045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 83216 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Cytoreduction Surgical Procedures; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment - Carboplatin, CRS, HIPEC (Experimental): Beginning 4-8 weeks after completion of chemotherapy, patients undergo CRS. Patients then receive carboplatin IP over 90 minutes immediately following CRS.
  Interventions: Drug: Carboplatin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Cytoreductive Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV and IP
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Cytoreductive Surgery — Undergo CRS
  Other Names: Operation; Surgery; Surgical; Surgical Interventions; Surgical Procedure; Surgical Procedures

SUMMARY:
This phase II trial studies how well hyperthermic intraperitoneal chemotherapy works in improving quality of life in patients with stage IIIC-IV ovarian, fallopian tube, or primary peritoneal cancer. In hyperthermic intraperitoneal chemotherapy, the chemotherapy is warmed before being used and may help the drugs get into the cancer cells better, minimize the toxicity of the drugs on normal cells, and help to kill any cancer cells left over after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe quality of life in patients with advanced ovarian cancer treated with standard of care (SOC) neoadjuvant chemotherapy (NAC) followed by cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) at 6 weeks post-treatment.

SECONDARY OBJECTIVES:

I. To describe quality of life in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC at 3 and 6 months post-treatment.

II. To describe neurotoxicity in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC.

III. To describe abdominal discomfort in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC.

IV. To describe toxicities in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC.

V. To describe the response rate in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC.

VI. To describe progression-free survival (PFS) in patients with advanced ovarian cancer treated with NAC followed by CRS with HIPEC.

OUTLINE: Beginning 4-8 weeks after completion of chemotherapy, patients undergo CRS. Patients then receive carboplatin intraperitoneally (IP) over 90 minutes immediately following CRS.

After completion of chemotherapy, patients are followed up at 30 days, and 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-mucinous, epithelial stage 3 or 4 carcinoma of the ovary, fallopian tube or peritoneum.
* Patients must not have received treatment for another malignancy within 3 years of enrollment (patients who have received hormone therapy within 3 years of enrollment are still eligible).
* Patients must have received at least 3 but not more than 6 cycles of carboplatin-doublet based IV neoadjuvant chemotherapy and achieved at least stable disease (radiographically confirmed) at the conclusion of this therapy.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have adequate organ and marrow function as defined below (within 30 days of registration):
* Absolute neutrophil count >= 1,500/mcL (within 30 days of registration)
* Platelets >= 75,000/mcL (within 30 days of registration)
* Total bilirubin =< 1.5 mg/dL (within 30 days of registration)
* Creatinine clearance >= 50 mg/dL (within 30 days of registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional upper limit of normal (within 30 days of registration)
* Alkaline phosphatase =< 3 x institutional upper limit of normal (within 30 days of registration)
* The effects of HIPEC on the developing human fetus are unknown. For this reason, and because carboplatin doublet therapy consists of pregnancy category D agents, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with extra-abdominal metastatic disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin doublet agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because carboplatin doublet therapy consists of pregnancy category D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with carboplatin doublet therapy, breastfeeding should be discontinued.
* Men are excluded from participating due to the site specific nature of the disease being studied.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelly, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period was January 2019 through December 2023.
Period: Overall Study
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Started | 50
Completed | 23 (Completed the Month 12 (after surgery) visit)
Not Completed | 27
Not completed — Death | 3
Not completed — Withdrawal by Subject | 15
Not completed — Did not complete protocol treatment | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50
Tumor Location [Count of Participants; unit: Participants]
  Ovary | 33
  Peritoneum | 17

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (QOL) Assessed Using Functional Assessment of Cancer Therapy-Ovarian Questionnaire (FACT-O)
Description: This is a descriptive study. QOL will be measured using the Fact-O questionnaire and treated as a continuous outcome. The distribution of QOL at 6 weeks post-treatment will be examined. Descriptive statistics such as mean, standard deviation, median and interquartile range will be calculated.
  The FACT-O consists of 39 questions answered with five-point Likert Scales (0-4). The possible range of scores is 0-156, and higher scores indicate a better quality of life.
Time Frame: At 6 weeks post treatment
Population: All participants did not have data collected for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 30
score on a scale | 116.32 (25.37)

2. Secondary Outcome: Abdominal Discomfort Assessed Using Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Abdominal Discomfort Questionnaire
Description: To describe abdominal discomfort at up to 3 times points during the study, descriptive statistics will be calculated and presented based on a 4-item score from FACT-GOG/AD. Counts and percentages will be calculated. Mean and standard deviation also will be calculated. This approach will be treated as a sensitivity analysis.
  The Abdominal Discomfort section of the FACT-O uses 4 questions with five-point Likert Scales (0-4). The possible range of scores is 0-16, and higher scores indicate a better quality of life (less discomfort),
Time Frame: Pre-treatment (baseline), 3 months after surgery, 6 months after surgery
Population: The most patients completed the survey at 6 months after surgery; most of them also completed the survey at baseline, and the fewest completed the survey at 3 months after surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 48
score on a scale
  Pre-treatment: number analyzed (Participants) | 46
  Pre-treatment | 1.76 (2.7)
  3 months after surgery: number analyzed (Participants) | 22
  3 months after surgery | 1.79 (2.4)
  6 months after surgery | 3.13 (4.4)

3. Secondary Outcome: Number of Toxicities Reported (National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0)
Description: The toxicities will be measured by the number and severity of adverse events defined by CTCAE version 5.0. Counts and percentages will be calculated for each type of adverse event. The counts were grouped in the table below. A particular count might include several occurrences of the same event (eg, anemia) or one occurrence of several different events.
Time Frame: Up to 6 weeks post treatment
Population: All participants able to receive the full protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 41
Participants
  Non-Serious Adverse Events: Zero Adverse Events | 0
  Non-Serious Adverse Events: One to Four Adverse Events | 2
  Non-Serious Adverse Events: Five to Nine Adverse Events | 6
  Non-Serious Adverse Events: Ten to Fourteen Adverse Events | 13
  Non-Serious Adverse Events: Fifteen to Nineteen Adverse Events | 11
  Non-Serious Adverse Events: Twenty or More Adverse Events | 9
  Serious Adverse Events: Zero Adverse Events | 32
  Serious Adverse Events: One to Four Adverse Events | 6
  Serious Adverse Events: Five to Nine Adverse Events | 2
  Serious Adverse Events: Ten to Fourteen Adverse Events | 1
  Serious Adverse Events: Fifteen to Nineteen Adverse Events | 0
  Serious Adverse Events: Twenty or More Adverse Events | 0

4. Secondary Outcome: Neurotoxicity Assessed Using Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity Questionnaire
Description: Neurotoxicity at up to three time points in the study will be described. The neurotoxicity subscale is an 11-item measure from FACT/GOG-NTX. The possible range of scores is 0 to 44, with higher scores indicating lower quality of life (more neurotoxicity).
Time Frame: Up to 6 months
Population: 47 patients completed this survey at baseline, 27 at 6 weeks post-surgery, 22 at 3 months post-surgery and 19 at 6 months post-surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 47
score on a scale
  Baseline | 33.92 (8.7)
  6 weeks post surgery: number analyzed (Participants) | 27
  6 weeks post surgery | 33.51 (9.25)
  3 months post surgery: number analyzed (Participants) | 22
  3 months post surgery | 35.59 (8.61)
  6 months post surgery: number analyzed (Participants) | 19
  6 months post surgery | 33.38 (10.01)

5. Secondary Outcome: Progression Free Survival
Description: Progression free survival will be estimated using Kaplan-Meier methods, using the time from the study registration up to date of progression, date of last contact, or death, whichever comes first.
Time Frame: Up to 2 years from study enrollment
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 50
months | 12.46 [9.2 to 15.2]

6. Secondary Outcome: Quality of Life (QOL) Assessed Using Functional Assessment of Cancer Therapy-Ovarian (FACT-O)
Description: The distribution of QOL based on the Fact-O questionnaire at 3 months post-treatment will be examined. The descriptive statistics of QOL at 3 months post-treatment will be presented.
  The FACT-O consists of 39 questions answered with five-point Likert Scales (0-4). The possible range of scores is 0-156, and higher scores indicate a better quality of life.
Time Frame: At 3 months post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 22
score on a scale | 126.11 (20.25)

7. Secondary Outcome: Quality of Life (QOL) in Patients With Advanced Ovarian Cancer Assessed Using Functional Assessment of Cancer Therapy-Ovarian (FACT-O)
Description: The distribution of QOL based on the Fact-O questionnaire at 6 months post-treatment will be examined. The descriptive statistics of QOL at 6 months post-treatment will be presented.
  The FACT-O consists of 39 questions answered with five-point Likert Scales (0-4). The possible range of scores is 0-156, and higher scores indicate a better quality of life.
Time Frame: At 6 months post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 20
score on a scale | 119.53 (31.40)

8. Secondary Outcome: Response Rates Evaluated According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: The best overall response using RECIST criteria will be determined for each evaluable patient and proportions achieving a complete or partial response will be estimated with 95% confidence intervals. Complete response means all target lesions have disappeared; partial response requires at least a 30% decrease in the sum of the longest diameters of target lesions from baseline. Progressive disease is defined by a 20% increase in the sum of the longest diameters of target lesions or the appearance of new lesions. Stable disease is defined as the absence of sufficient changes to qualify for partial response or progressive disease.
Time Frame: Up to 6 weeks post surgery
Population: All participants who were able to complete all treatment according to protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
Number analyzed (Participants) | 41
Participants
  Complete Reponse | 17
  Partial Response | 17
  Stable Disease | 3
  Progressive Disease | 4

ADVERSE EVENTS:
Time Frame: Up to 1 year post-surgery.
Description: Adverse event data were recorded with each cycle of chemotherapy, at the post-surgery visit, and at 6 weeks, 3, 6 and 12 months post-surgery.
  Adverse events were recorded only for those who completed the full protocol treatment (n=41), but all enrolled patients (n=50) were following for mortality, since all enrolled patients were at risk for mortality.
Arm/Group | Treatment - Carboplatin, CRS, HIPEC
All-Cause Mortality (participants affected / at risk) | 6/50
Serious Adverse Events (participants affected / at risk) | 27/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Carboplatin, CRS, HIPEC (N=41)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Atelaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment - Carboplatin, CRS, HIPEC (N=41)
Anemia (Blood and lymphatic system disorders) | 38 (69)
Leukocytes (Blood and lymphatic system disorders) | 5 (6)
Sinus Tachycardia (Cardiac disorders) | 10 (10)
Abdominal Distension (Gastrointestinal disorders) | 4 (7)
Abdominal Pain (Gastrointestinal disorders) | 18 (21)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Ileus (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 18 (26)
Vomiting (Gastrointestinal disorders) | 18 (20)
Chills (General disorders) | 4 (4)
Limb Edema (General disorders) | 6 (7)
Fatigue (General disorders) | 26 (38)
Pain (General disorders) | 7 (8)
Urinary Tract Infection (Infections and infestations) | 4 (5)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (10)
Alkaline phosphatase increased (Investigations) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 7 (8)
Lymphocyte count decreased (Investigations) | 25 (37)
Metabolic Acidosis (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 13 (17)
Platelet count decreased (Investigations) | 27 (48)
White blood cell decreased (Investigations) | 22 (39)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 35 (59)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 30 (41)
Hypokalemia (Metabolism and nutrition disorders) | 24 (35)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (13)
Hyponatremia (Metabolism and nutrition disorders) | 20 (32)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 8 (10)
Headache (Nervous system disorders) | 5 (5)
Paresthesia (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hypertension (Vascular disorders) | 12 (21)
Hypotension (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03188432/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03188432/ICF_000.pdf